CLINICAL TRIAL: NCT05425355
Title: INTACT-HIP: INTravenous Acetaminophen vs. Oral Randomized Controlled Trial in HIP Fracture Patients - a Feasibility Trial
Brief Title: Intravenous vs Oral Acetaminophen in Postoperative Hip Fracture Adult Patients
Acronym: INTACT-HIP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jean Wong, Associate Professor, University of Toronto, Department of Anesthesiology and Pain Medicine, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-5733
Record Dates: First submitted 2022-05-16; First posted 2022-06-21 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Hip-fracture; Surgery
Keywords: elderly; acetaminophen; oral vs intravenous; hip fracture surgery
MeSH Terms: conditions — Hip Fractures | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: The study intervention will start after the surgery for the hip fracture with administration of the study drugs, starting in the post-anesthesia care unit (PACU). All patients will receive both a tablet and an IV solution every 6 hours for 48 hours, for a total of 8 doses. In the intravenous (IV) group, the IV study drug will be IV acetaminophen and the oral study drug will be a placebo tablet; vice versa, in the per oral (PO) group, the IV study drug will be normal saline and the pill will be acetaminophen. After 48 hours, all the patients will receive oral acetaminophen every 6 hours as per usual practice
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous (IV) acetaminophen plus oral placebo (Experimental): In this group, the IV study drug will be IV acetaminophen and the oral study drug will be a placebo tablet.
  Interventions: Drug: Intravenous (IV) acetaminophen + oral placebo
- Intravenous (IV) placebo plus oral acetaminophen (Active Comparator): In this group the IV study drug will be normal saline and the pill will be acetaminophen
  Interventions: Drug: Intravenous (IV) placebo plus oral acetaminophen

INTERVENTIONS:
Drug: Intravenous (IV) acetaminophen + oral placebo — Postoperatively patients will receive both a tablet and an IV solution every 6 hours for 48 hours, for a total of 8 doses. In this group, the IV study drug will be IV acetaminophen and the oral study drug will be a placebo tablet.
  Arms: Intravenous (IV) acetaminophen plus oral placebo
Drug: Intravenous (IV) placebo plus oral acetaminophen — Postoperatively patients will receive both a tablet and an IV solution every 6 hours for 48 hours, for a total of 8 doses. In this group the IV study drug will be normal saline and the pill will be acetaminophen
  Arms: Intravenous (IV) placebo plus oral acetaminophen

SUMMARY:
The INTACT-HIP trial study will evaluate feasibility of conducting a randomized, double-blinded controlled trial comparing postoperative treatment with intravenous (IV) acetaminophen versus oral acetaminophen, in older adults undergoing hip fracture surgery.

The results of this feasibility trial will be used to inform designing a larger, multi-center, randomized controlled trial to assess the efficacy of IV acetaminophen compared to oral acetaminophen to reduce delirium and improve other clinical and patient-centered outcomes after hip fracture surgery. It will randomize 42 older adults to receive either oral or IV acetaminophen after hip fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age and older
* Patients who were ambulating without human assistance before fracture, with any type of non-neoplastic hip fracture
* Patients undergoing surgical treatment as an inpatient

Exclusion Criteria:

* Patients with neoplastic hip fracture
* Severe cognitive impairment (Montreal Cognitive Assessment (MoCA) <10)
* Pre-existing delirium
* Known hypersensitivity or allergy to acetaminophen
* Severe or chronic liver or kidney dysfunction
* Planned postoperative ventilation
* Swallowing issues and/or dysphagia
* English language limitation
* Weight <50kg

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Trial feasibility-Recruitment | 30 days
  Feasibility as assessed by recruitment rate. This will be assesses as proportion of patients enrolled in the study compared to the number of patients meeting the inclusion/exclusion criteria.
Trial feasibility-Attrition | 30 days
  Feasibility as assessed by attrition rates. This will be defined as the proportion of patients completing the study at follow-up compared to the enrolled patients.
Trial feasibility-Availability of human resources | 30 days
  Feasibility as assessed by lack of availability of human resources). Inability to include patient in study due to lack of pharmacist or research assistant availability will be documented.
Trial feasibility-Comply study procedures | 30 days
  Feasibility as assessed by failure to comply with study procedures. Failure to provide study drug at scheduled time will be documented.
Trial safety | 30 days
  Safety will be assessed as the number of participants experiencing intervention-related adverse or serious adverse events.

SECONDARY OUTCOMES:
Postoperative pain | Before surgery, on day of surgery, and days 1,2,3 after surgery
  Pain will be assessed using the visual analogue (VAS) scale (0-10) at rest and movement, with 0=no pain and 10=worst pain possible
Opioid consumption | Before surgery, on day of surgery, and days 1,2,3 after surgery
  Oral morphine equivalents (OMEQS) in milligrams
Delirium | On day of surgery, and days 1,2, 3 after surgery
  Delirium incidence will be measured using the Confusion assessment method (CAM)-Long Form
Cognitive dysfunction | Before surgery and day 3 after surgery (or at discharge time if hospital stay less than 3 days after surgery)
  Cognitive dysfunction will be assessed using the Montreal Cognitive Assessment (MoCA)
Overall health and disability | Baseline and at 30 days after surgery
  Overall health and disability will be measured using the WHO Disability Assessment Schedule, version 2.0 (WHODAS 2.0), a 12-item validated measure that assesses cognition, mobility, self-care, interpersonal relationships, work and household roles, and participation in society
Depression screen | Before surgery and day 3 after surgery (or at discharge time if hospital stay less than 3 days after surgery)
  Patient Health Questionnaire (PHQ)-2 a 2-question questionnaire will be used as a validated measure to screen for depression.
Ambulation | Before surgery and day 3 after surgery (or at discharge time if hospital stay less than 3 days after surgery)
  Ambulation will be assessed as the ability to walk 10 feet or across a room without human assistance
Post-operative adverse events | On day of surgery, days 1,2, 3 after surgery, and at 30 days after surgery
  Post-operative adverse events will be obtained from the study institution's National Surgical Quality Improvement Project (NSQIP) database as as death, ICU admission, standardized cardiac, respiratory and neurological postoperative events, and readmission to hospital.
Discharge location | At the time of discharge (at 1-3 days after surgery in most cases)
  Location of discharge after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean Wong, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital (UHN), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jahr JS, Breitmeyer JB, Pan C, Royal MA, Ang RY. Safety and efficacy of intravenous acetaminophen in the elderly after major orthopedic surgery: subset data analysis from 3, randomized, placebo-controlled trials. Am J Ther. 2012 Mar;19(2):66-75. doi: 10.1097/MJT.0b013e3182456810. PMID 22354127
- [Result] Chen DX, Yang L, Ding L, Li SY, Qi YN, Li Q. Perioperative outcomes in geriatric patients undergoing hip fracture surgery with different anesthesia techniques: A systematic review and meta-analysis. Medicine (Baltimore). 2019 Dec;98(49):e18220. doi: 10.1097/MD.0000000000018220. PMID 31804347
- [Result] Harris MJ, Brovman EY, Urman RD. Clinical predictors of postoperative delirium, functional status, and mortality in geriatric patients undergoing non-elective surgery for hip fracture. J Clin Anesth. 2019 Dec;58:61-71. doi: 10.1016/j.jclinane.2019.05.010. Epub 2019 May 14. PMID 31100691